CLINICAL TRIAL: NCT06369870
Title: Interpectoral-pectoserratus Plane Block for Minimally Invasive Aortic Valve Replacement Via Right Anterior Minithoracotomy: a Single Centre, Prospective, Double-blind, Randomized Controlled Superiority Trial
Brief Title: Interpectoral-pectoserratus Plane Block for Minimally Invasive Aortic Valve Replacement Via Right Anterior Minithoracotomy
Acronym: PAINCARE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Bart Vaes, MD, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAINCARE
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Analgesic Effect
Keywords: interpectoral-pectoserratus plane block; aortic valve replacement via right anterior minithoracotomy; IPP-PSP block; AVR-RAT
MeSH Terms: interventions — Levobupivacaine; Sodium Chloride; Control Groups

STUDY DESIGN:
Intervention Model Description: The trial is designed as a single-center, prospective, double-blind, randomized controlled superiority trial. Patients will be randomly assigned to either the IPP-PSP block group or the sham block group (placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant, anesthesiologist, study nurse, surgeon, nor the doctors and nurses in the Intensive Care Unit will know the participant's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levobupivacaine Hydrochloride 0.25 % Injectable Solution (Active Comparator): Unilateral (right) IPP-PSP block with 30 mL levobupivacaine 0.25%, administered after the closure of the wounds. After wound closure, the IPP-PSP block is performed at the level of the 4th rib. At the pre-axillary line, the pectoralis major, the pectoralis minor and the serratus anterior muscle are identified. At first, the needle is positioned in the fascial plane between the pectoralis minor and the serratus anterior muscle. The needle position is confirmed by hydro-dissection of this plane with 2 mL of normal saline 0.9%.The 20 ml syringe with trial drug solution is injected in this pectoserratus plane (PSP). The needle tip is repositioned in the interpectoral plane between both the pectoralis major and minor muscle. The 10 ml syringe with trial drug solution is administered in this interpectoral plane (IPP).
  Interventions: Drug: Levobupivacaine Hydrochloride 0.25 % Injectable Solution
- Sodium chloride 0.9% (Sham Comparator): Unilateral (right) IPP-PSP block with 30 mL normal saline 0.9%, administered after the closure of the wounds. Unilateral (right) IPP-PSP block with 30 mL normal saline 0.9%, administered after the closure of the wounds. The IPP-PSP block procedure will be carried out as described in the Active Comparator.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Levobupivacaine Hydrochloride 0.25 % Injectable Solution — After wound closure, the IPP-PSP block is performed at the level of the 4th rib. At the pre-axillary line, the pectoralis major, the pectoralis minor and the serratus anterior muscle are identified. At first, the needle is positioned in the fascial plane between the pectoralis minor and the serratus anterior muscle. The needle position is confirmed by hydro-dissection of this plane with 2 mL of normal saline 0.9%.The 20 ml syringe with trial drug solution is injected in this pectoserratus plane (PSP). The needle tip is repositioned in the interpectoral plane between both the pectoralis major and minor muscle. The 10 ml syringe with trial drug solution is administered in this interpectoral plane (IPP).
  Other Names: IPP-PSP block; Intervention group
  Arms: Levobupivacaine Hydrochloride 0.25 % Injectable Solution
Drug: Sodium chloride 0.9% — Unilateral (right) IPP-PSP block with 30 mL normal saline 0.9%, administered after the closure of the wounds. The IPP-PSP block procedure will be carried out as described in the intervention description of the IPP-PSP block.
  Other Names: Sham block; Control group
  Arms: Sodium chloride 0.9%

SUMMARY:
The goal of this clinical trial is to evaluate the analgesic effect of locoregional anaesthesia, specifically the interpectoral pectoserratus plane (IPP-PSP) block, in comparison to a placebo (sham block) after Aortic Valve Replacement via Right Anterior Minithoracotomy (AVR-RAT). The main question the trial aims to answer is: Can the IPP-PSP block effectively reduce opioid consumption within the first 48 hours after AVR-RAT surgery? The purpose is to understand the impact of the IPP-PSP block on postoperative pain. Therefore, the aim is to investigate the influence of the IPP-PSP block on the amount of pain medication administered during the patients' first 48 hours after surgery.

Participants, who are scheduled for AVR-RAT surgery, will be randomly assigned to receive either the IPP-PSP block or the sham block. Researchers will compare opioid consumption among other outcomes, including differences in pain scores, incidence of nausea and vomiting, quality of recovery, quality of life, and the length of hospital stay between the two groups.

Patients will be monitored during their hospitalization, and a follow-up phone call will be conducted 30 days after surgery.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the analgesic effect of an interpectoral-pectoserratus plane (IPP-PSP) block compared to a placebo (sham block) in patients undergoing aortic valve replacement via right anterior minithoracotomy (AVR-RAT). The primary objective is to determine whether the IPP-PSP block effectively reduces opioid consumption during the first 28 hours post-surgery.

The trial is designed as a single-center, prospective, double-blind, randomized controlled superiority trial. It will enroll adult patients aged 18 years or older who are scheduled for minimally invasive AVR-RAT and meet specific inclusion criteria. Exclusion criteria are established to ensure the safety and integrity of the trial.

Patients undergoing minimally invasive AVR-RAT will be randomly assigned to either the IPP-PSP block group or the sham block group.

The primary endpoint of the trial is the cumulative opioid consumption (in oral morphine milligram equivalents (OMEs)) within the first 48 postoperative hours after completion of the surgical procedure. Secondary outcomes include the number of episodes of postoperative pain, time to need for rescue medication, incidence of respiratory complications, PaCO2 levels, postsurgical recovery, episodes of postoperative nausea and vomiting, time to extubation in the Intensive Care Unit (ICU), ICU length of stay, hospital length of stay, quality of life, number of days alive and at home after surgery, and vital status at 30 days post-operative.

The trial aims to enroll a total of 144 patients, with 72 patients randomized into each group. Blinding will be implemented, meaning neither the participant, anesthesiologist, study nurse, surgeon, nor the doctors and nurses in the Intensive Care Unit will know the participant's group assignment.

The anesthesia and monitoring proceed as usual for such procedures. After the anesthesiologist administered the IPP-PSP block or a placebo at the end of the procedure, the participant will be transferred to the ICU. During the hospital stay, they will be regularly asked to assess their pain level, and additional pain relief will be administered, if necessary.

To assess quality of recovery and quality of life differences between groups, participants will complete two questionnaires the day before surgery. A recovery questionnaire will be completed at three time points post-surgery (day 1, day 2, and day 7 after the surgery). Participants will be involved in the trial for a total of 31 days, with follow-up during hospitalization and a follow-up phone call 30 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older);
* Patients scheduled for minimally invasive aortic valve replacement via right anterior minithoracotomy;
* Patients with American Society of Anesthesiologists (ASA) physical status classification II, III or IV;
* Patients with European System for Cardiac Operative Risk Evaluation (EuroSCORE) 2 ≤ 4%;
* Patient has given written, free and informed consent.

Exclusion Criteria:

* BMI > 35;
* Patients under legal protection (curatorship, guardianship);
* Patients subject to a legal protection measure;
* An adult who is incapable or unable to give consent;
* Patients requiring emergency surgery within 24 hours;
* Chronic opioid use (> 3 administrations per week or continuous transdermal therapy, longer than the last 3 months);
* Patients known with chronic pain;
* Patients known with an allergy to levobupivacaine or drugs used as standard of care, including amongst others piritramide, dexamethasone, propofol, remifentanil, rocuronium, acetaminophen, ondansetron;
* Patients who receive medication that could possibly interact with levobupivacaine (mexiletine, ketoconazole, theophylline);
* Patients who took monoamine oxidase (MAO) inhibitors within the last 2 weeks before surgery;
* Patients with chronic renal failure (dialysis dependent, estimated glomerular filtration rate (eGFR) < 30 ml.min-1.(1,73 m²)-1) ;
* Patients with severe hepatic impairment (Model for End-Stage Liver Disease (MELD) score ≥ 20);
* Patients with preoperative cognitive dysfunction (Mini Mental State Examination (MMSE) score < 24);
* Patients with uncontrolled epilepsy;
* Patients with severe arterial hypotension (Systolic Arterial Pressure (SAP) < 90 mmHg, cardiogenic shock);
* Patients who simultaneously participate in another interventional clinical trial;
* Soft tissue infection in the area of the procedure;
* Patients who are pregnant, parturient or breast-feeding women;
* Patients who are unable to sufficiently speak and write in the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption | in the first 48 hours after completion of the surgical procedure
  Cumulative opioid consumption (in oral morphine milligram equivalents (OMEs)) in the first 48 postoperative hours after the completion of the surgical procedure

SECONDARY OUTCOMES:
Number of episodes of postoperative pain | In the first 48 hours after completion of the surgical procedure
  Number of episodes of postoperative pain (NRS score ≥ 4) at rest and at deep inspiration in the first 48 postoperative hours after the completion of the surgical procedure
Time to need for rescue medication | In the first 48 hours after completion of the surgical procedure
  Time to need for rescue medication for breakthrough pain (e.g. tramadol, oxycodone) in the first 48 postoperative hours after the completion of the surgical procedure (minutes)
Number of patients with respiratory complications | During hospital stay (on average 7 days)
  Number of patients with respiratory complications, leading to non-invasive ventilation (NIV) or high-flow nasal cannula (HFNC) oxygen therapy, orotracheal intubation for more than 24 hours or orotracheal re-intubation
PaCO2 levels | During the 48 postoperative hours after the completion of the surgical procedure or until Intensive Care Unit (ICU) discharge, whichever occurs first;
  Levels of arterial partial pressure of carbon dioxide (PaCO2) measured every 4 hours during the 48 postoperative hours after the completion of the surgical procedure or until Intensive Care Unit (ICU) discharge, whichever occurs first
Postsurgical Quality of Recovery measured by the Quality of Recovery questionnaire | Day before, first, second and seventh day after surgery
  Postsurgical recovery by Quality of Recovery questionnaire (QoR-15NL) on day before (D-1), first (D1), second (D2) and seventh (D7) day after surgery.
  The minimum score on the Quality of Recovery questionnaire is 0 and the maximum score 150. Higher scores mean better quality of recovery.
Number of episodes of postoperative nausea and vomiting | Number of episodes of postoperative nausea and vomiting (PONV) in the first 48 postoperative hours after the completion of the surgical procedure: nausea yes/no, vomiting: yes/no
  Number of episodes of postoperative nausea and vomiting (PONV) in the first 48 postoperative hours after the completion of the surgical procedure: nausea yes/no, vomiting: yes/no
Time to extubation | Minutes (assessed up to 6 hours after surgery)
  Time to extubation of the patient in the Intensive Care Unit
Number of hours spent in the Intensive Care Unit | Hours (on average 48 hours)
  Number of hours spent in the Intensive Care Unit (until ready for discharge)
Hospitalization duration | Days (on average 7 days)
  Number of days in the hospital between surgery and first hospital discharge
Quality of life measured by the 5 level version of the EuroQoL-5 Dimension questionnaire | Day before and 30 days after surgery
  The quality of life by the EQ-5D-5L questionnaire on the day before surgery and 30 days (D30) after surgery.
  The minimum health utility value of the Belgian EQ-5D-5L value set is -0.532 and the maximum value 1 in Belgium. Higher utility scores mean better health related quality of life.
Days alive and at home | 30 (+7) days after surgery
  Number of days alive and at home after surgery (DAH30)
Vital status (whether the patient is alive or dead) | 30 (+7) days after surgery
  Vital status at 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bart Vaes, MD, Principal Investigator — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ Maria Middelares, Ghent, East-Flanders, Belgium